CLINICAL TRIAL: NCT03089541
Title: Electronic Cigarette Use in Young Adult Men and Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: APT Foundation, Inc. (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1612018726; 1P50DA036151-01 (NIH)
Record Dates: First submitted 2017-03-20; First posted 2017-03-24 (Actual); Results first posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Cigarette Smoking; Tobacco Use
MeSH Terms: conditions — Cigarette Smoking; Tobacco Use

STUDY DESIGN:
Intervention Model Description: 30 non-treatment seeking young adult e-cigarette/cigarette dual users (15 males/15 females) will participate in a contingency-management reinforced 1 week observation period
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Survey Arm (Experimental): Will receive incentives for completing surveys and evidence of tobacco use status daily for 1 week
  Interventions: Behavioral: Survey Arm

INTERVENTIONS:
Behavioral: Survey Arm — Contingency Management for completion of surveys and evidence of tobacco use status

SUMMARY:
This one-year pilot study of 30 non-treatment seeking young adult e-cigarette/combustible tobacco product dual users (15 males/15 females) will use smartphone-based ecological momentary assessment (EMA) to gather real-time data of e-cigarette and combustible tobacco product behaviors during a 1-week cigarette/e-cigarette dual use period .(1) Participants will respond to daily random prompts assessing in-the-moment use of e-cigarettes/cigarettes and the subjective factors (ratings of satisfaction and withdrawal) and contextual factors (location, activity, social cues) associated with each episode of use. Participants will also complete daily electronic diaries to document e-cigarette use episodes/day, and satisfaction with the e-cigarette experience during the study.

ELIGIBILITY:
Inclusion Criteria:

1. be 18 through 29 years of age;
2. Smoke cigarettes;
3. have experience with e-cigarette use;
4. fluent in English;
5. have a functioning cell phone for personal use ;
6. have access to wireless networks at least once daily;
7. have self-reported good health.

Exclusion Criteria.

1. report serious medical illness;
2. are women who are currently/planning to be pregnant or breastfeeding.

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2018-02-16 (Actual); Primary Completion 2018-10-17 (Actual); Study Completion 2018-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deepa R Camenga, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Camenga DR, Haeny AM, Krishnan-Sarin S, O'Malley SS, Bold KW. Pilot Ecological Momentary Assessment Study of Subjective and Contextual Factors Surrounding E-Cigarette and Combustible Tobacco Product Use among Young Adults. Int J Environ Res Public Health. 2021 Oct 20;18(21):11005. doi: 10.3390/ijerph182111005. PMID 34769525

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through flyers, targeted advertisements on Facebook, Instagram, Craigslist, public boards in local colleges, and through the university research volunteer database.
Period: Overall Study
Arm/Group | Survey Arm
Started | 29
Completed | 29
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Survey Arm
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.9 (3.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 14
  More than one race | 2
  Unknown or Not Reported | 10
Region of Enrollment [Number; unit: participants]
  United States | 29
Highest Level of Education Completed [Count of Participants; unit: Participants]
  High School | 18
  Some College/College | 11
Baseline FTCD Score [Mean (Standard Deviation); unit: units on a scale] — The Fagerström Test for Nicotine Dependence is a standard instrument for assessing the intensity of physical addiction to nicotine. The six-item instrument provides ordinal measure of nicotine dependence related to cigarette smoking. In scoring the FTND, yes/no items are scored from 0 to 1 and multiple-choice items are scored from 0 to 3. The items are summed to yield a total score of 0-10. The higher the total Fag xscore, the more intense is the patient's physical dependence on nicotine.
  units on a scale | 2.6 (2.4)
E-cigarette Device Type Used [Count of Participants; unit: Participants]
  Cartridge | 12
  Tank | 12
  Mod | 2
  Other | 3
Cigarettes Smoked/Day [Count of Participants; unit: Participants]
  Non-Daily | 9
  1 to 5 | 10
  6 to 10 | 3
  10 to 20 | 6
  21+ | 1
Type of Combustible Tobacco Product Used in Past Week [Count of Participants; unit: Participants]
  Cigarettes Only | 21
  Cigarette + Hookah | 3
  Cigarettes + Cigars | 2
  Cigarettes + Cigars + Hookah | 3

OUTCOME MEASURES:

1. Primary Outcome: Contextual Factors Associated With Tobacco Use Episode Reported Via Ecological Momentary Assessment
Description: Participant responses to prompt during ecological momentary assessment about their activity, location, and companionship during a tobacco use episode that occurred within the past 15 minutes.
Time Frame: week 1
Population: non-treatment seeking young adults who use both e-cigarettes and combustible tobacco products
Measure: Number; unit: tobacco use episodes
Units Other Than Participants: tobacco use episodes
Groups:
- E-cigarette Use Episode: Episode of e-cigarette use reported via ecological momentary assessement
- Episode of Combustible Tobacco Product Use: Episode of Combustible Tobacco Product Use reported via ecological momentary assessment.
Arm/Group | E-cigarette Use Episode | Episode of Combustible Tobacco Product Use
Number analyzed (Participants) | 29 | 29
Number analyzed (tobacco use episodes) | 68 | 111
tobacco use episodes
  Eating/Drinking | 3 | 22
  Working/Reading/Studying | 11 | 12
  Traveling | 5 | 3
  Socializing | 15 | 18
  In a public space | 34 | 83
  Alone | 45 | 33
Statistical Analysis 1: Comparison: E-cigarette Use Episode vs Episode of Combustible Tobacco Product Use; Comparison on Eating/Drinking using a model adjusted for timing of the assessment (weekend, time of day (am vs. pm), and day of study (1 to 7). The significance level was 0.05; Test type: Superiority; p = 0.002, Regression, Logistic; Odds Ratio (OR) = 0.17, 95% CI 2-sided [0.06 to 0.52]
Statistical Analysis 2: Comparison: E-cigarette Use Episode vs Episode of Combustible Tobacco Product Use; Comparison on Traveling using a model adjusted for timing of the assessment (weekend, time of day (am vs. pm), and day of study (1 to 7)). The significance level was 0.05; Test type: Superiority; p = 0.07, Regression, Logistic; Odds Ratio (OR) = 2.65, 95% CI 2-sided [0.92 to 7.65]
Statistical Analysis 3: Comparison: E-cigarette Use Episode vs Episode of Combustible Tobacco Product Use; Comparison on Working/Reading/Studying using a model adjusted for timing of the assessment (weekend, time of day (am vs. pm), and day of study (1 to 7). The significance level was 0.05; Test type: Superiority; p = 0.40, Regression, Logistic; Odds Ratio (OR) = 1.46, 95% CI 2-sided [0.59 to 3.64]
Statistical Analysis 4: Comparison: E-cigarette Use Episode vs Episode of Combustible Tobacco Product Use; Comparison on Socializing using a model adjusted for timing of the assessment (weekend, time of day (am vs. pm), and day of study (1 to 7). The significance level was 0.05; Test type: Superiority; p = 0.60, Regression, Logistic; Odds Ratio (OR) = 1.34, 95% CI 2-sided [0.51 to 3.53]
Statistical Analysis 5: Comparison: E-cigarette Use Episode vs Episode of Combustible Tobacco Product Use; Model on Public Space adjusted for timing of the assessment (weekend, time of day (am vs. pm), and day of study (1 to 7)). The significance level was 0.05; Test type: Superiority; p = 0.06, Regression, Logistic; Odds Ratio (OR) = 1.80, 95% CI 2-sided [0.96 to 3.38]

ADVERSE EVENTS:
Time Frame: 1 week
Arm/Group | Survey Arm
All-Cause Mortality (participants affected / at risk) | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 0/29

LIMITATIONS AND CAVEATS:
Small sample

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-10-18): https://cdn.clinicaltrials.gov/large-docs/41/NCT03089541/Prot_SAP_000.pdf
  • Informed Consent Form (2018-09-07): https://cdn.clinicaltrials.gov/large-docs/41/NCT03089541/ICF_001.pdf